CLINICAL TRIAL: NCT05984862
Title: Bandage Versus No-Bandage After Follicular Unit Extraction Hair Transplantation
Brief Title: Role of Bandage After FUE Hair Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pak Medical and Diagnostic Center (Other)
Responsible Party: Principal Investigator, Muhammad Sarfraz Khan, Research Associate, Pak Medical and Diagnostic Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PMDC-23-07-6745
Record Dates: First submitted 2023-07-25; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Hair Loss/Baldness
Keywords: Hair Loss; Follicular Unit Extraction; Hair transplantation; Wound healing
MeSH Terms: conditions — Alopecia | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: This is a single center, triple-blind, within subject split scalp study investigating the comparison of bandage versus no bandage donor site post FUE. Twenty-five subjects desiring to undergo FUE for hair restoration will have bandage on one half of the donor area on the back of the scalp and no-bandage on the other side for 24 hours post procedure. The sides of the scalp will be randomized, and the evaluating physician will be blinded. Subjects will be evaluated, photographed, and will fill out subject reported questionnaires live at days 1 (+1) and 7 (±1) post procedure.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized, triple-blind, split-scalp study. The subjects will know what side of the scalp the bandage products are applied. However, during evaluation, the subjects and analyst will be shown close-up pictures of the two sides without exposing the patient's identity and actual sides.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Treatment left (Experimental): A randomized side of the scalp will be covered with bandage, the other side with no bandage.
  Intervention: Device: Treatment - Bandage
  Interventions: Device: Bandage
- Experimental: Treatment right (Experimental): A randomized side of the scalp will be covered with bandage, the other side with no bandage.
  Intervention: Device: Treatment - Bandage
  Interventions: Device: Bandage

INTERVENTIONS:
Device: Bandage — To determine if using bandage versus no-bandage, plays a role in limiting severity and duration of signs and symptoms of acute inflammation post follicular harvesting procedure
  Other Names: wound healing

SUMMARY:
The aim of this interventional study is to determine the role of bandage on the follicular donor sites on the scalp after FUE hair transplantation.

A randomized side of the scalp will be covered using bandage, the other side will be left naked. Subjects under study will be evaluated after the procedure is completed, and day 1 and day 7 post-procedure during the healing phase. This will in turn help, answering the importance of bandage in healing of the donor site post-hair transplantation.

DETAILED DESCRIPTION:
In this modern era, hair-transplantation has become very common. Interests in wound healing is not new; with every passing day, different techniques are introduced to get better results for the patients. The current literature available online shows that many hair-transplant centers have stated about using bandage on the donor area post-transplantation, however, there isn't a single study available to augment this use of bandage. On the other hand, data regarding application of antibiotic ointments and silicon gels is available. The punctures made during FUE are only of 9-10mm, requiring no sutures. In addition to this, the blood supply of the scalp also favors quick healing. The process of re-epithelization starts within a few hours of injury and progresses over the first 1 to 3 days. Most of the clinics remove, the bandage after 24hrs, disrupting the healing process of the skin. In the present study, the investigators sought to compare bandage versus no-Bandage donor site in terms of healing. The investigators hypothesize that, compared with bandage site, no-bandage donor site after FUE will have reduce post-procedural downtime and donor site inflammation ultimately, enhancing patient satisfaction with the procedure. The long-term goal of this study is to get evidence-based usage of bandage, if results are in contrast with the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Able to provide informed consent
* Planning to undergo follicular unit extraction hair restoration

Exclusion Criteria:

* Significant medical or surgical conditions
* Unable to give informed consent
* Immunocompromised

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Wound healing change over time from day 0 to day +1 (+1), to day +7 (±1) | duration of the study be evaluated and rated on days 1 (+1) and 7 (±1) post procedure for both the bandage and no bandage sites
  Bandage has protection role to some extent; however, removal of bandage will affect the normal healing of donor site. Healing Response (4-point ordinal scale) LEFT SIDE
  * Not healed at all (0%)
  * Mildly healed (33%)
  * Moderately healed (66%)
  * Completely healed (100%)
  RIGHT SIDE
  * Not healed at all (0%)
  * Mild healing (33%)
  * Moderately healed (66%)
  * Completely healed (100%)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sarfraz Khan, BSc, MBBS, Study Director — Pak Medical and Diagnostic Center

IPD SHARING:
Plan to Share IPD: No